CLINICAL TRIAL: NCT03315377
Title: Lunatocapitate Fusion Versus Four-corner Fusion for SNAC and SLAC Arthritis. A Randomized Comparison.
Brief Title: Lunatocapitate Fusion Versus Four-corner Fusion for SNAC and SLAC Arthritis.
Acronym: MIKA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Thorsten Schriever, MD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIKA1
Record Dates: First submitted 2017-08-21; First posted 2017-10-20 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Wrist Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lunate-Capitate Fusion (LCF) (Active Comparator): Operation with a Lunate-Capitate Fusion (LCF) for SLAC or SNAC arthritis.
  Interventions: Procedure: Lunate-Capitate Fusion (LCF)
- Four Corner Fusion (4CF) (Active Comparator): Operation with a Four Corner Fusion (4CF) for SLAC or SNAC arthritis
  Interventions: Procedure: Four Corner Fusion (4CF)

INTERVENTIONS:
Procedure: Lunate-Capitate Fusion (LCF) — Operation with lunate-capitate-fusion (LCF)
  Arms: Lunate-Capitate Fusion (LCF)
Procedure: Four Corner Fusion (4CF) — Operation with four-corner-fusion (4CF)
  Arms: Four Corner Fusion (4CF)

SUMMARY:
Hypothesis: Lunate-capitate-fusion (LCF) results in comparable outcome (i.e. not worse) to four-corner-fusion (4CF) for Scaphoid Nonunion Advanced Collapse (SNAC) and Scapholunate Advanced Collapse (SLAC) arthritis regarding functional results (grip strength).

Design: Prospective randomised comparison. Inclusion criteria: SNAC or SLAC arthritis requiring a salvage procedure (grade 2-3).

Exclusion criteria: SNAC or SLAC arthritis grade 4 (panarthritis). Inability to co-operate with the follow-up protocol (language difficulties, severe psychiatric disorder or drug addiction).

DETAILED DESCRIPTION:
Surgical method:

Patient will be operated in axially plexus with a dorsal approach through the 3d and 4th extensor tendon compartments. The wrist joint capsule will be opened with a Berger incision. After excision of the scaphoid and preparation of the articular surfaces to be fused, the bones will be fixated with k-wires. Bone autograft from the scaphoid, crista or radius will be used according to the surgeon's preference based on the condition of the fusion surfaces. The wrist be immobilized in a short arm plaster cast until the fusions are radiologically healed after10-12 weeks. The k-wires will be extracted in local anesthesia after another 2-6 weeks.

Sample size:

This study will have a power of 80% to show that the mean grip strength for LC fusion is as least as high as the mean for 4CF (non-inferiority). This assumes that the means for the LC fusion and the 4CF are equal (at 70% of the uninjured side) with a common within-group standard deviation of 14 (Salzman et al. 2015), that a difference of 10% or less is unimportant, that the sample size in the two groups will be 25 and 25, and the alpha (1 tailed) is set at 0,05.Formally, the null hypothesis is that the mean for lunocapitate fusion is 10% lower than the mean for 4CF, and that the study has power of 80,1% to reject this null. Equivalently, the likelihood is 80,1% that the 95% confidence interval for the mean difference will exclude a difference of 10% in favor of 4CF.

We aim to include 60 patients to cover for a certain loss to follow-up.

Assessment:

Patients will be assessed regarding range of motion and grip strength and complete the DASH and PRWE questionnaires before surgery (baseline) and 1 and 2 years postoperatively.

Radiology:

Plain anterior and lateral radiographs will be obtained 1 and 2 years postoperatively for purpose of the study. According to the standard treatment protocol, clinical and radiological healing assessment will be conducted 10-12 weeks postoperatively. Radiographs will be analyzed by a radiologist.

Complications will be recorded 1 and 2 years postoperatively.

Analyzes:

The Mann-Whitney and Chi-square tests will be used for non-parametric data (DASH, PRWE and presence of arthritis and complications). T-test will be used for numerical data (ROM, grip strength).

ELIGIBILITY:
Inclusion Criteria:

- SNAC or SLAC arthritis grade 2-3

Exclusion Criteria:

* SNAC or SLAC arthritis grade 4
* Inability to cooperate with the follow-up protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Grip strength | 1 year postoperatively
  Hand grip strength measured with Jamar dynamometer

SECONDARY OUTCOMES:
DASH score | 1 year postoperatively
  Disability of the Arm, Hand and Shoulder (DASH) questionnaire
PRWE score | 1 year postoperatively
  Patient Rated Wrist Evaluation (PRWE)
Range of motion (ROM) | 1 year postoperatively
  Wrist ROM measured with a goniometer
EQ5D (for analysis of health economy) | 1 year postoperatively
  Quality of life questionnaire
Complications | 1 year postoperatively
  Infection, nonunion
Progress of arthritis | 1 year postoperatively
  Radiological signs of radiocarpal arthritis on CT scans

CONTACTS AND LOCATIONS:
Overall Officials: Maria Wilcke, MD, PhD, Study Director — Stockholm, Sweden
Locations (1):
- Dept of Handsurgery SÖS, Stockholm, Sweden